CLINICAL TRIAL: NCT00005577
Title: A PEDIATRIC PHASE I STUDY OF GEMCITABINE (NSC# 613327) IN SOLID TUMORS
Brief Title: Gemcitabine in Treating Children With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02246; CCG-0954; CDR0000064886 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-05-02; First posted 2004-04-02 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2002-12

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Gemcitabine

ARMS (1):
- Arm I (Experimental): Patients receive gemcitabine IV over 30 minutes weekly for 2 weeks. Patients achieving objective response or stable disease after 3 weeks may receive additional courses of therapy every 3 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of gemcitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity.
  Interventions: Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: gemcitabine hydrochloride

SUMMARY:
Phase I trial to study the effectiveness of gemcitabine in treating children who have refractory solid tumors. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Estimate the maximum tolerated dose of gemcitabine in children and adolescents with refractory solid tumors.

II. Assess the toxicity of gemcitabine in this patient population. III. Determine the pharmacokinetic profile of gemcitabine in male and female children and adolescents.

IV. Assess the antitumor activity of gemcitabine within a phase I study.

OUTLINE: This is a dose escalation study.

Patients receive gemcitabine IV over 30 minutes weekly for 2 weeks. Patients achieving objective response or stable disease after 3 weeks may receive additional courses of therapy every 3 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of gemcitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity. Patients are followed at week 4 and then every 6 months until death.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant solid tumor Confirmation made at original diagnosis
* No bone marrow involvement
* Refractory to conventional therapy and other therapies of higher priority according to CCG Phase I/II Priority List

PATIENT CHARACTERISTICS:

* Age: 1 to 21
* Performance status: 0-2
* Life expectancy: At least 2 months
* Absolute neutrophil count at least 1,000/mm3
* Platelet count at least 100,000/mm3 (transfusion independent)
* Hemoglobin at least 10 g/dL (transfusions allowed)
* Bilirubin no greater than 1.5 times normal
* AST less than 2.5 times normal
* Creatinine no greater than 1.5 times normal OR creatinine clearance or radioisotope GFR at least 70 mL/min
* No seizure disorder Not pregnant or nursing
* Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior cytokine therapy and recovered
* No prior bone marrow transplantation
* No more than 3 prior combination or single agent chemotherapy regimens
* At least 3 weeks since prior chemotherapy (6 weeks since nitrosoureas) and recovered

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 1996-08; Primary Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John S. Holcenberg, MD, Study Chair — Seattle Children's Hospital
Locations (23):
- United States (22):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Cancer Center and Beckman Research Institute, City of Hope, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia